CLINICAL TRIAL: NCT01461213
Title: An Open Label Dose Escalation Phase 1 Clinical Trial of Retinal Gene Therapy for Choroideraemia Using an Adeno-associated Viral Vector (AAV2) Encoding Rab-escort Protein 1 (REP1)
Brief Title: Gene Therapy for Blindness Caused by Choroideremia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); University College, London (Other); Manchester University NHS Foundation Trust (Other Government); University of Manchester (Other); University Hospital Southampton NHS Foundation Trust (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHM09/01; 2009-014617-27 (EudraCT Number)
Record Dates: First submitted 2011-10-21; First posted 2011-10-28 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Choroideremia
Keywords: Tapetoretinal degeneration, choroideraemia, X-linked; retinitis pigmentosa
MeSH Terms: conditions — Choroideremia; Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose 1 (Experimental): Dose 1 = single subretinal injection of vector suspension containing approximately 10e10 rAAV2.REP1 genome particles. Six patients have now received Dose 1.
  Interventions: Drug: rAAV2.REP1
- Dose 2 (Experimental): Dose 2 = single subretinal injection of vector suspension containing approximately 10e11 rAAV2.REP1 genome particles. Three patients thus far have received Dose 2.
  Interventions: Drug: rAAV2.REP1

INTERVENTIONS:
Drug: rAAV2.REP1 — Single subretinal injection of rAAV2.REP1 vector suspension containing 10e12 genome particles per ml. Dose 1 = dose containing approximately 10e10 rAAV2.REP1 genome particles. Dose 2 = dose containing approximately 10e11 rAAV2.REP1 genome particles.
  Other Names: Adeno-associated viral vector

SUMMARY:
- Primary objective: To assess the safety and tolerability of the AAV.REP1 vector, administered at two different doses to the retina in 12 patients with a diagnosis of choroideremia.

- Secondary Objective: To identify any therapeutic benefit as evidenced by a slowing down of the retinal degeneration assessed by functional and anatomical methods in the treated eye compared to the control eye 24 months after gene delivery.

DETAILED DESCRIPTION:
Detailed description may be found in the following scientific publication:

Retinal gene therapy in patients with choroideremia: initial findings from a phase 1/2 clinical trial, The Lancet, Volume 383, Issue 9923, Pages 1129 - 1137 (29 March 2014).

Links: www.thelancet.com/journals/lancet/article/PIIS0140-6736(13)62117-0/abstract ; http://dx.doi.org/doi:10.1016/S0140-6736(13)62117-0

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study,
* Male aged 18 years or above,
* Diagnosed with choroideraemia and in good health,
* Active disease with SLO changes visible within the macula region,
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study,
* Vision at least 6/60 or better in the study eye.

Exclusion Criteria:

* Female and child participants (under the age of 18),
* Men unwilling to use barrier contraception methods, if relevant,
* Previous history of retinal surgery or ocular inflammatory disease (uveitis),
* Grossly asymmetrical disease or other ocular morbidity which might confound use of the fellow eye as a long-term control,
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study,
* Participants who have participated in another research study involving an investigational product in the previous 12 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months
  Best corrected visual acuity, following cataract surgery if indicated

SECONDARY OUTCOMES:
Microperimetry, OCT and fundus autofluorescence | 24 months
  Structure function correlations at the margins of the retinal degeneration

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MacLaren, MB ChB DPhil, Study Chair — University of Oxford, Oxford Radcliffe Hospitals NHS Trust and Moorfields Eye Hospital; Miguel C Seabra, MD PhD, Principal Investigator — Imperial College London; Andrew R Webster, MD, Principal Investigator — UCL Institute of Ophthalmology and Moorfields Eye Hospital; Susan M Downes, MD, Principal Investigator — Oxford University Hospitals NHS Trust; Graeme C Black, MB BCh DPhil, Principal Investigator — University of Manchester and Central Manchester University Hospitals NHS Foundation Trust; Andrew J Lotery, MD, Principal Investigator — University of Southampton and Southampton University Hospitals Trust; Len W Seymour, PhD, Principal Investigator — University of Oxford; Tanya Tolmachova, PhD, Principal Investigator — Imperial College London
Locations (4):
- United Kingdom (4):
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - St Mary's Hospital, Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Oxford Radcliffe Hospitals NHS Trust, Oxford
  - Eye Unit, Southampton University Hospitals NHS Trust, Southampton

REFERENCES:
- [Derived] Simunovic MP, Jolly JK, Xue K, Edwards TL, Groppe M, Downes SM, MacLaren RE. The Spectrum of CHM Gene Mutations in Choroideremia and Their Relationship to Clinical Phenotype. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6033-6039. doi: 10.1167/iovs.16-20230. PMID 27820636
- [Derived] Xue K, Oldani M, Jolly JK, Edwards TL, Groppe M, Downes SM, MacLaren RE. Correlation of Optical Coherence Tomography and Autofluorescence in the Outer Retina and Choroid of Patients With Choroideremia. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(8):3674-84. doi: 10.1167/iovs.15-18364. PMID 27403996
- [Derived] Seitz IP, Zhour A, Kohl S, Llavona P, Peter T, Wilhelm B, Zrenner E, Ueffing M, Bartz-Schmidt KU, Fischer MD. Multimodal assessment of choroideremia patients defines pre-treatment characteristics. Graefes Arch Clin Exp Ophthalmol. 2015 Dec;253(12):2143-50. doi: 10.1007/s00417-015-2976-4. Epub 2015 Mar 7. PMID 25744334
- [Derived] MacLaren RE, Groppe M, Barnard AR, Cottriall CL, Tolmachova T, Seymour L, Clark KR, During MJ, Cremers FP, Black GC, Lotery AJ, Downes SM, Webster AR, Seabra MC. Retinal gene therapy in patients with choroideremia: initial findings from a phase 1/2 clinical trial. Lancet. 2014 Mar 29;383(9923):1129-37. doi: 10.1016/S0140-6736(13)62117-0. Epub 2014 Jan 16. PMID 24439297